CLINICAL TRIAL: NCT02743767
Title: Frequency of Airway Complications During General Anaesthesia After Introducing Five Handling Adaptations
Acronym: Papaya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PAPAYA
Record Dates: First submitted 2016-04-05; First posted 2016-04-19 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Airway Complications
Keywords: Airway management; General anaesthesia; Critical incidents; Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Before interventions (No Intervention): Only observational activity for this arm, to record the frequency and triggering factors of airway complications during general anaesthesia.
- After interventions (Experimental): After introducing five different treating adaptations in airway management we want to record the frequency of airway complications during general anaesthesia.
  Interventions: Procedure: Introducing five different treating adaptations

INTERVENTIONS:
Procedure: Introducing five different treating adaptations — Immediate Bag-valve mask ventilation after administering of muscle relaxants, optimized preoxygenation, introducing of a preinterventional checklist, increased usage of video laryngoscopy and immediate hand alternately if frustrated intubation.
  Arms: After interventions

SUMMARY:
The purpose of this study is to determine if five simple adaptations in airway management of patients undergoing general anaesthesia can reduce minor and major airway complications.

After a first detection of causes of airway complications during general anaesthesia investigators initiated five different interventions in airway management, which were: immediate bag-valve mask ventilation after administering of muscle relaxants, optimized preoxygenation, introducing of a preinterventional checklist, increased usage of video laryngoscopy and immediate change of provider in case of failed intubation.

In a second phase of this observational study investigators want to evaluate if these five interventions can reduce minor and major airway complications during general anaesthesia.

Additionally, investigators want to record how many critical incidents (CIRS) occur during this observational period and how many of them will be reported by the involved stuff.

ELIGIBILITY:
Inclusion Criteria:

* Must receive a general anaesthesia with any form of airway management

Exclusion Criteria:

* Anaesthesia without airway management
* Patients who do not give or who withdraw general consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7455 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Reduction of airway complications after introducing five treatment adaptations | 2 months

SECONDARY OUTCOMES:
Postoperative side effects after routinely general anaesthesia | 2 months
Frequency of reporting critical incident (CIRS) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD MME FERC, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Huber M, Greif R, Pedersen TH, Theiler L, Kleine-Brueggeney M. Risk patterns of consecutive adverse events in airway management: a Bayesian network analysis. Br J Anaesth. 2023 Mar;130(3):368-378. doi: 10.1016/j.bja.2022.11.007. Epub 2022 Dec 22. PMID 36564247
- [Derived] Pedersen TH, Ueltschi F, Hornshaw T, Greif R, Theiler L, Huber M, Kleine-Brueggeney M. Optimisation of airway management strategies: a prospective before-and-after study on events related to airway management. Br J Anaesth. 2021 Nov;127(5):798-806. doi: 10.1016/j.bja.2021.07.030. Epub 2021 Sep 15. PMID 34535275